CLINICAL TRIAL: NCT01514890
Title: Cohort of Therapeutic Failure and Resistances in Patients Treated With a Protease Inhibitor (Telaprevir or Boceprevir), Pegylated Interferon (PEG-IFN) and Ribavirin (RBV) Included in the French Early Access Program for the Use of Protease Inhibitors in Genotype 1 Patients Who Failed to Eradicate HCV With a Previous Standard PEG-IFN and RBV Combination.
Brief Title: French Cohort of Therapeutic Failure and Resistances in Patients Treated With a Protease Inhibitor (Telaprevir or Boceprevir), Pegylated Interferon and Ribavirin
Acronym: CUPIC
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS CO20; 2010-A01273-36 (Other: AFSSAPS)
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Telaprevir
- Boceprevir

SUMMARY:
The purpose fo the study is to evaluate the efficacy defined by the sustained virological response (SVR), in patients with compensated cirrhosis treated with PEG-IFN, RBV and telaprevir or boceprevir in the French Early Access Program for the use of protease inhibitors or after the approval of these drugs through the the marketing authorization.

DETAILED DESCRIPTION:
Methodology: Multicentric French national cohort with prospective collection of data and constitution of biobank, in HCV genotype 1 patients with compensated cirrhosis who failed to eradicate HCV with the combination PEG-IFN and RBV, treated with protease inhibitor (telaprevir or boceprevir), PEG-IFN and RBV, included in the French Early Access Program for the use of protease inhibitors or after approval of these drugs through the the marketing authorization.

Primary objective: Evaluate the efficacy defined by the sustained virological response (SVR), in patients with compensated cirrhosis treated with PEG-IFN, RBV and telaprevir or boceprevir in the French Early Access Program for the use of protease inhibitors or after the approval of these drugs.

Estimated enrollment: 900 patients treated in the French Early Access Program for the use of protease inhibitors and after the marketing authorization approval.

Treatments:

* with telaprevir: triple combination with PEG-IFN alfa-2a, 180 µg/week, ribavirin 1000 to 1200 mg/d according the body weight and telaprevir 750 mg/8h, for 12 weeks followed by PEG-IFN and RBV for 36 weeks for a total duration of treatment of 48 weeks.
* or with boceprevir: triple combination with PEG-IFN alfa-2b, 1,5 µg/kg/week, RBV 800 to 1400 mg/d according the body weight and boceprevir 800 mg/8h. The treatment will begin after a lead in phase of PEG-IFN and RBV for 4 weeks, followed by a triple combination (PEG-IFN, RBV and boceprevir)during 44 weeks for a total duration of treatment of 48 weeks.

Estimated planning:

* study start date: February 2011
* enrollment period: 14 months
* subject participation duration: 12 months of treatment and 12 months of follow-up = 24 months
* total study duration: 38 months. The last visit of the last enrolled patient is prevised in February 2014, the end of analysis on biobank in May 2014 (long term follow up of resistant mutants).

Some blood samples will be preserved for scientific future research.

Study design: national French multicentric cohort in patients with HCV-related cirrhosis treated in the French Early Access Program for the use of boceprevir or telaprevir or after the marketing authorization approval of these drugs associated with PEG-IFN and RBV with a collection of clinical and biological data and constitution of a biobank.

ELIGIBILITY:
Inclusion Criteria:

* patients who need the criteria of French Early Access Program for boceprevir and telaprevir or after the marketing authorization approval:

  * patients aged of 18 years or more with chronic hepatitis C
  * relapsers or partial-responders or null-responders to treatment with PEG'IFN α2a or 2b associated or not with RBV
  * chronic infection with genotype 1 HCV
  * fibrosis Metavir score of 4 (cirrhosis)
  * without decompensated liver disease
  * naïve of direct anti-viral treatment
  * without HIV or HBV co-infection
* signature of participation to the cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C in genotype 1 Who Failed to Eradicate HCV With a Previous Standard PEG-IFN and RBV Combination
Sampling Method: Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Rate of sustained virological response (SVR) defined by an undetectable RNA by real-time PCR. | 6 months after discontinuation of therapy (at week 72)

SECONDARY OUTCOMES:
Virological response during and after the treatment with determination of HCV RNA levels as prevised by the French Early Access Program for the use of protease inhibitors and after the approval. | at D0, W4, W8, W12, W24, W48 and 12 (W60) and 24 (W72) weeks after the discontinuation of treatment
  This will allow to define:
  * rate of non response (detectable RNA during the treatment)
  * rate of virological breakthrough (undetectable HCV RNA then detectable during the treatment)
  * rate of virological relapse after the discontinuation of treatment (undetectable HCV RNA at the end of therapy then detectable after the treatment)
early viral kinetic | at the D0, W1, W2 and W4
Rate of premature discontinuation of protease inhibitor, RBV and/or PEG-IFN | in may 2014 (3 month after study completion date)
occurrence of resistant mutants in partial responders (detectable RNA) or after the occurrence of virological breakthrough and long term evolution of these mutations (on serum bank) | in may 2014 (3 month after study completion date)
Evolution of quality of life scores | in may 2014 (3 month after study completion date)
Evaluation of therapeutic observance with auto-questionnaires | in may 2014 (3 month after study completion date)
Rate of adaptation of dosage of protease inhibitors, RBV and/or PEG-IFN | in may 2014 (3 month after study completion date)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe HEZODE, Principal Investigator — GHU H. Mondor; Fabrice CARRAT, Methodologist, Study Chair — Unité INSERM 707
Locations (1):
- Hôpital Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Sultanik P, Mallet V, Lagaye S, Casrouge A, Dorival C, Barthe Y, Fontaine H, Hezode C, Mottez E, Bronowicki JP, Carrat F, Theodorou I, Abel L, Gayat E, Fontanet A, Pol S, Albert ML; ANRS CO20-CUPIC. Plasma apolipoprotein H limits HCV replication and associates with response to NS3 protease inhibitors-based therapy. Liver Int. 2015 Jul;35(7):1833-44. doi: 10.1111/liv.12759. Epub 2015 Jan 23. PMID 25556540
- [Derived] Hezode C, Fontaine H, Dorival C, Zoulim F, Larrey D, Canva V, De Ledinghen V, Poynard T, Samuel D, Bourliere M, Alric L, Raabe JJ, Zarski JP, Marcellin P, Riachi G, Bernard PH, Loustaud-Ratti V, Chazouilleres O, Abergel A, Guyader D, Metivier S, Tran A, Di Martino V, Causse X, Dao T, Lucidarme D, Portal I, Cacoub P, Gournay J, Grando-Lemaire V, Hillon P, Attali P, Fontanges T, Rosa I, Petrov-Sanchez V, Barthe Y, Pawlotsky JM, Pol S, Carrat F, Bronowicki JP; CUPIC Study Group. Effectiveness of telaprevir or boceprevir in treatment-experienced patients with HCV genotype 1 infection and cirrhosis. Gastroenterology. 2014 Jul;147(1):132-142.e4. doi: 10.1053/j.gastro.2014.03.051. Epub 2014 Apr 3. PMID 24704719
- [Derived] Hezode C, Fontaine H, Dorival C, Larrey D, Zoulim F, Canva V, de Ledinghen V, Poynard T, Samuel D, Bourliere M, Zarski JP, Raabe JJ, Alric L, Marcellin P, Riachi G, Bernard PH, Loustaud-Ratti V, Metivier S, Tran A, Serfaty L, Abergel A, Causse X, Di Martino V, Guyader D, Lucidarme D, Grando-Lemaire V, Hillon P, Feray C, Dao T, Cacoub P, Rosa I, Attali P, Petrov-Sanchez V, Barthe Y, Pawlotsky JM, Pol S, Carrat F, Bronowicki JP; CUPIC Study Group. Triple therapy in treatment-experienced patients with HCV-cirrhosis in a multicentre cohort of the French Early Access Programme (ANRS CO20-CUPIC) - NCT01514890. J Hepatol. 2013 Sep;59(3):434-41. doi: 10.1016/j.jhep.2013.04.035. Epub 2013 May 10. PMID 23669289